CLINICAL TRIAL: NCT01376245
Title: A 24-week Study to Evaluate the Efficacy and Safety of Fluticasone Furoate/Vilanterol Inhalation Powder Delivered Once Daily Via a Dry Powder Inhaler Compared With Placebo in Subjects of Asian Ancestry With Chronic Obstructive Pulmonary Disease
Brief Title: A 24-week Study of Fluticasone Furoate/Vilanterol Inhalation Powder in Subjects of Asian Ancestry With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113684
Record Dates: First submitted 2011-06-09; First posted 2011-06-20 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone furoate/vilanterol (Experimental): Inhaled corticosteroid/long acting beta-agonist
  Interventions: Drug: fluticasone furoate/vilanterol
- placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fluticasone furoate/vilanterol — Inhaled corticosteroid/long acting beta-agonist
  Arms: fluticasone furoate/vilanterol
Drug: Placebo — matching placebo
  Arms: placebo

SUMMARY:
The purpose of the study is to investigate the efficacy and safety of fluticasone furoate/vilanterol Inhalation Powder compared with placebo over a 24 weeks treatment period in subjects of Asian ancestry with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis define by ATS(American Thoracic Society)/ ERS (European Respiratory Society)
* Subjects of Asian ancestry
* Valid informed consent
* Current or former smoker
* > or = 2 on the modified Medical Research Council Dyspnea Scale at Screening

Exclusion Criteria:

* Pregnancy
* A current diagnosis of asthma
* alpha1-antitrypsin deficiency as the underlying cause for COPD
* Other active, respiratory disorders
* Have lung volume reduction surgery within 12 months prior to Screening
* A chest X-ray or CT (Computerised Tomography) scan reveals evidence of clinical significant abnormalities not believed to be due to the presence of COPD
* Poorly controlled COPD: acute worsening of COPD managed by corticosteroids, antibiotics, or treatments prescribed by a physician 6 weeks prior to Screening, or requires hospitalisation due to poorly controlled COPD 12 weeks prior to Screening
* Lower respiratory tract infection requires antibiotics within 4 weeks prior to Screening
* Other disease or abnormalities, in the opinion of the investigator, would put the safety of the subject at risk during the study or would affect safety or efficacy analysis if the disease/condition exacerbated during the study
* Subject with carcinoma that has not been in complete remission for at least 5 years, carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded if the subject has been considered cured within 5 years since diagnosis.
* Subject has a history of hypersensitivity to any of the study medications or components of the inhalation powder. Subject has a history of severe milk protein allergy that, in the opinion of the investigator, contraindicates the subject's participation will also be excluded.
* Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years prior to Screening
* Subjects who are medically unable to withhold albuterol, ipratropium for 4 hrs and/or theophylline for 12 hrs prior to spirometry testing.
* Subjects use a list of prohibited medications specified in the study protocol, including but not limited to traditional or herbal medications for the treatment of COPD
* Subject requires long-term oxygen therapy or nocturnal oxygen therapy for greater than 12 hours a day
* Pulmonary rehabilitation: subjects who are in the maintenance phase are not excluded.
* Non-compliance
* Questionable validity of the Informed Consent
* Prior use of study medication or other investigational drugs
* Affiliation with investigator site

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- China (12):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanning, Guangxi
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- GSK Investigational Site, Quezon City, Philippines
- South Korea (3):
  - GSK Investigational Site, Jeonju-si, Jeollabuk-Do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Gyeonggi-do
- Taiwan (5):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan County

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Zheng J, de Guia T, Wang-Jairaj J, Newlands AH, Wang C, Crim C, Zhong N. Efficacy and safety of fluticasone furoate/vilanterol (50/25 mcg; 100/25 mcg; 200/25 mcg) in Asian patients with chronic obstructive pulmonary disease: a randomized placebo-controlled trial. Curr Med Res Opin. 2015 Jun;31(6):1191-200. doi: 10.1185/03007995.2015.1036016. PMID 25830381
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113684 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants (par.) completed a 2-week Run-in Period for symptom scores at baseline and to establish a stable baseline. Par. were then randomized to a 24-week (wk) Treatment Period. 880 par. were screened, 744 entered the RIP and 646 par were randomized, out of which 643 par received >=1 study treatment dose.
Groups:
- Placebo- Run-in: Participants received placebo once daily (OD) in the morning for 2 weeks. In addition, participants were provided supplemental albuterol/salbutamol (metered dose inhaler [MDI] or nebules) to be used as needed throughout the study.
- Placebo: Participants received placebo once daily (OD) in the morning for 24 weeks. In addition, participants were provided supplemental albuterol/salbutamol (metered dose inhaler [MDI] or nebules) to be used as needed throughout the study.
- FF /VI 50/25 µg OD: Participants received Fluticasone Furoate (FF)/Vilanterol (VI) 50/25 micrograms (µg) OD in the morning over the 24-week treatment period. In addition, participants were provided albuterol/salbutamol (MDI or nebules) to be used as needed throughout the study.
- FF/VI 100/25 µg OD: Participants received FF/VI 100/25 µg OD in the morning over the 24-week treatment period. In addition, participants were provided albuterol/salbutamol (MDI or nebules) to be used as needed throughout the study.
- FF/VI 200/25 µg OD: Participants received FF/VI 200/25 µg OD in the morning over the 24-week treatment period. In addition, participants were provided albuterol/salbutamol (MDI or nebules) to be used as needed throughout the study.
Period: 2-wk Single-blind Placebo Run-in Period
Arm/Group | Placebo- Run-in | Placebo | FF /VI 50/25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Started | 744 | 0 | 0 | 0 | 0
Completed | 643 | 0 | 0 | 0 | 0
Not Completed | 101 | 0 | 0 | 0 | 0
Not completed — Did Not Meet Continuation Criteria | 66 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 28 | 0 | 0 | 0 | 0
Period: 24-week, Double-blind Treatment Period
Arm/Group | Placebo- Run-in | Placebo | FF /VI 50/25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Started | 0 | 162 | 160 | 161 | 160
Completed | 0 | 130 | 135 | 138 | 134
Not Completed | 0 | 32 | 25 | 23 | 26
Not completed — Adverse Event | 0 | 16 | 7 | 8 | 18
Not completed — Lack of Efficacy | 0 | 4 | 5 | 4 | 3
Not completed — Protocol Violation | 0 | 2 | 0 | 2 | 1
Not completed — Met Protocol-Defined Stopping Criteria | 0 | 2 | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 6 | 9 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF /VI 50/25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | Total
Number analyzed (Participants) | 162 | 160 | 161 | 160 | 643
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (8.78) | 65.2 (8.41) | 65.1 (9.19) | 62.7 (8.65) | 64.4 (8.80)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 16 | 12 | 15 | 59
  Male | 146 | 144 | 149 | 145 | 584
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 151 | 149 | 150 | 148 | 598
  Asian - South East Asian | 11 | 11 | 11 | 12 | 45

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Clinic Visit Pre-dose Trough FEV1 at Day 169
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 was defined as the pre-dose and pre-bronchodilator FEV1, which was obtained at each clinic visit. Baseline is defined as the mean of the two assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1.Trough FEV1 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing at each clinic visit. Change from Baseline was calculated as the average at each clinic visit minus the Baseline value. Analysis was performed using a repeated measures model with covariates of treatment, smoking status at screening (stratum), baseline - mean of the two assessments made 30 minutes pre-dose and immediately pre-dose on Day 1, day, day by baseline and day by treatment interactions.
Time Frame: Baseline to Day 169
Population: Intent-to-Treat (ITT) Population: all randomized par. who received at least one dose of study medication. Number of par. presented represents those with data available at the time point being presented, however, all par. in the ITT population without missing covariate information with at least one post BL measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- FF/VI 50/25 µg OD: Participants received Fluticasone Furoate (FF)/Vilanterol (VI) 50/25 micrograms (µg) OD in the morning over the 24-week treatment period. In addition, participants were provided albuterol/salbutamol (MDI or nebules) to be used as needed throughout the study.
Arm/Group | Placebo | FF/VI 50/25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 126 | 134 | 136 | 131
Liters | -0.027 (0.0184) | 0.113 (0.0183) | 0.152 (0.0181) | 0.167 (0.0182)
Statistical Analysis 1: Comparison: Placebo vs FF/VI 50/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted Maximum Likelihood (REML)-based repeated measures approach (MMRM); Least Squares Mean Difference = 0.140, 95% CI 2-sided [0.089 to 0.191]
Statistical Analysis 2: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted Maximum Likelihood (REML)-based repeated measures approach (MMRM); Least Squares Mean Difference = 0.179, 95% CI 2-sided [0.129 to 0.230]
Statistical Analysis 3: Comparison: Placebo vs FF/VI 200/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted Maximum Likelihood (REML)-based repeated measures approach (MMRM); Least Squares Mean Difference = 0.194, 95% CI 2-sided [0.143 to 0.245]

2. Secondary Outcome: Mean Change From Baseline in Chronic Respiratory Disease Questionnaire Self-administered Standardized (CRQ-SAS) Dyspnea Domain Score at Day 168
Description: CRQ-SAS measures 4 domains (fatigue, emotional function, mastery and dyspnea) of functioning of participants (par.) with COPD: mastery (amount of control the par. feels he/she has over COPD symptoms); fatigue (how tired the par. feels); emotional function (how anxious/depressed the par. feels); and dyspnea (how short of breath the par. feels during physical activities). Each domain is calculated separately and measured on a scale of 1-7 (1=maximum impairment; 7=no impairment). Dyspnea domain score is the mean of all non-missing responses for that domain. Only the dyspnea domain was measured as a secondary outcome. BL scores are the derived scores for each domain and total at Day 1 pre-dose. Change from BL was calculated as the average of the Day 168 values minus the BL value. Analysis performed used a repeated measures model with covariates of treatment, smoking status at screening (stratum), BL (derived scores at Day 1 pre-dose), day, day by BL, and day by treatment interactions.
Time Frame: Baseline (BL) and Day 168
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF/VI 50/25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 128 | 134 | 136 | 132
Scores on a scale | 0.09 (0.081) | 0.30 (0.080) | 0.43 (0.079) | 0.37 (0.080)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study medication to the end of treatment (up to Week 24).
Description: An on-treatment AE or SAE is defined as an AE with an onset on or after the start date of study medication, but not later than one day after the last date of study medication. SAEs and AEs were collected in members of the ITT Population, comprised of all participants randomized to treatment, who received at least one dose of the study medication.
Groups:
- FF/VI 50/25 µg OD: articipants received Fluticasone Furoate (FF)/Vilanterol (VI) 50/25 micrograms (µg) OD in the morning over the 24-week treatment period. In addition, participants were provided albuterol/salbutamol (MDI or nebules) to be used as needed throughout the study.
Arm/Group | Placebo | FF/VI 50/25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Serious Adverse Events (participants affected / at risk) | 14/162 | 9/160 | 7/161 | 14/160
Other Adverse Events (participants affected / at risk) | 27/162 | 33/160 | 34/161 | 40/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=162) | FF/VI 50/25 µg OD (N=160) | FF/VI 100/25 µg OD (N=161) | FF/VI 200/25 µg OD (N=160)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 3 | 8
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 2 | 0 | 2
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Renal embolism (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal infarct (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=162) | FF/VI 50/25 µg OD (N=160) | FF/VI 100/25 µg OD (N=161) | FF/VI 200/25 µg OD (N=160)
Upper respiratory tract infection (Infections and infestations) | 15 | 16 | 19 | 14
Nasopharyngitis (Infections and infestations) | 7 | 13 | 9 | 19
Pyrexia (General disorders) | 5 | 3 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6 | 3
Hypertension (Vascular disorders) | 1 | 1 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.